CLINICAL TRIAL: NCT02249572
Title: Vestibular Schwannoma - Radiosurgery or Expectation
Brief Title: Vestibular Schwannoma - Radiosurgery or Expectation: V-REX.
Acronym: V-REX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014/314
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Vestibular Schwannoma
Keywords: Vestibular schwannoma; Radiosurgery; Neurosurgery; Randomized
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: Block randomization of 100 individuals to radiosurgery or expectative treatment of vestibular schwannoma.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study investigator masked to whether patient has had radiosurgery og no active treatment. Scars due to radiosurgery frame hidden With surgical cap at all study consultations in all pts. Radiologist measuring tumor size masked as to treatment
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gamma knife radiosurgery (Experimental): Single fraction gamma knife radiosurgery given at 12 Gy to tumor periphery for vestibular schwannoma
  Interventions: Radiation: gamma knife radiosurgery
- Expectation (No Intervention): No active treatment given for vestibular schwannoma

INTERVENTIONS:
Radiation: gamma knife radiosurgery — Leksell Perfection model gamma knife.
  Arms: gamma knife radiosurgery

SUMMARY:
The purpose of this study is to compare the outcome of patients with vestibular schwannomas in two groups of randomised to either radiosurgery or expectation.

The optimal treatment for a small vestibular schwannoma is a matter of controversy and there are no class 1 studies investigating this. Even the natural tumor growth rate remains controversial and is reported to be from near 100% of cases showing growth to 40-60% in various reports. The clinical results of various treatment strategies are documented, but comparative studies are very few. Immediate radiosurgery or wait-and scan with subsequent treatment upon growth are two strategies that have both been used in many different centers. There are only two studies comparing these treatment modalities .These studies indicate significant effect of GKRS in reducing tumor growth, with less differences in hearing and complaint outcomes. None of the studies are blinded or randomised, allowing for bias.

The present study aims at comparing the two modalities above. To achieve this, we intend to randomise patients with newly diagnosed VS to either of Wait-and Scan or immediate radiosurgery.

The primary study endpoint is the relative tumor size measured as the ratio between tumor volume at four years compared with volume at inclusion. Secondary endpoints include symptom and sign development measured by clinical examination and by patient's responses to standardised validated questionnaires. In addition, the health economics involved with both strategies will be evaluated and compared, as well as the patient's working status.

Patients will be asked to participate if their VS is diagnosed within the last six months, their age is between 18 and 70, and pending there are no exclusion criteria (see below). A power analysis indicates that about 50 patients per group is sufficient.

In case of failure to recruit patients, we will change the design to a study based on patient's own choice of treatment.

The study will be announced according to international guidelines. A steering committee will monitor the study and an intermediate analysis will be performed when the study group has been followed for two years. If the effect aim is already observed, the study should nonetheless continue, as it is too early to evaluate the results after such a short time course.

It will also be discussed to do a follow-up of all patients ten years after inclusion.

DETAILED DESCRIPTION:
Study design and purpose:

Design: Randomised study blinded to observer on primary endpoint (tumor volume). Intention-to-treat, ie patients who cross over from conservative to GKRS group during the study period are assigned to their original group. Patients who refrain from radiosurgery despite randomisation are assigned to radiosurgery group.

Purpose: compare the treatment of small and medium-sized VS treated with a standardised dose of 12 Gy to the tumor periphery with expectative treatment.

Primary endpoint:

Growth measured as volume ratio V4years/Vbaseline and 1/volume doubling time, evaluated by T1 contrast MRI volumetry at one, two, three and four years.

Secondary endpoints:

Hearing acuity according to Gardner Robertson scale at four years (safety endpoint).

Conversion to other treatment during study period Adverse effects

Subjective complaints assessed by questionnaires:

Penn Vestibular Schwannoma QOL Scale EQ-50 Scale

Investigations:

Prior to inclusion: MRI less than 6 months showing VS.

After inclusion and at 1,2 3,4 years, all at study site:

MRI of inner ear (acoustic neuroma protocol) Balance platform Nystagmometry Audiometry

Effect registration:

Main variable:

Tumor volume, measured on a T1 contrast MRI scan with 2mm slice interval/thickness. For study, the measurement is to be done by a blinded observer.

Economy. Costs associated with study are financed by research donations from Helse-Vest and The National Center for Vestibular Schwannomas.

Radiology: Image based tumor volumes As the primary endpoint is relative tumor size, an accurate measure of tumor volume and changes thereof, is mandatory. This will be obtained using a state-of-the-art magnetic resonance imaging (MRI) system suited for acquiring high resolution (1mm3), three dimensional (3D) anatomical images. A 1.5T imaging system which meets the required field homogeneity will be used for imaging. The image contrast will be T1 weighted with gadolinium based contrast agent, yet a T2 weighted image volume will also be included (preferably also acquired in 3D). An identical imaging protocol will be acquired at each time point (prior to randomization, on site follow up, 4-year annual follow up), and image slices will be positioned according to anatomical landmarks in each patients to minimize variability across time. All 3D acquisitions will be performed with sagittal slicing to minimize artifacts, but will also be reformatted into coronal and axial views (1mm slice thickness, no gap between slices) on the scanner system.

The subsequent imaging processing, i.e. the estimation of tumor volume and longitudinal changes thereof, will be performed using available software at time of analysis.

Study schedule

Clinical examination, MRI, Questionnaires, Audiometry, Vestibular tests are done at baseline and then annually for 4 years. Patients randomised for radiosurgery are treated within 3 months after baseline.

ELIGIBILITY:
Inclusion Criteria:

* Vestibular schwannoma diagnosed by MRI of less than 6 months.
* Diameter 4-20mm. Willing to participate. Age 18 -70 years.

Exclusion Criteria:

* Dementia
* Active malignant disease
* Type II neurofibromatosis in patient or first grade relative.
* Other severe co-morbidity
* Type 2 neurofibromatosis in patient or first-grade relative

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Relative Tumor volume | 4 years
  Growth measured as volume ratio V4years/Vbaseline and 1/volume doubling time

SECONDARY OUTCOMES:
Hearing acuity | 4 years
  Hearing acuity according to Gardner Robertson scale at four years
Conversion to other treatment during study period | 4 years
  If patient is in need of other treatment for tumor (radiosurgery, microsurgery, other) within the time frame of the study
Subjective complaints | 4 years
  Penn Vestibular Schwannoma QOL Scale (PANQOL) EQ-50 Scale

OTHER OUTCOMES:
Neurovestibular testing | 4 years
  Outcomes of caloric test and Balance Platform test (Equitest, SOT)

CONTACTS AND LOCATIONS:
Overall Officials: Morten Lund-Johansen, MD PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Haukeland Unviersity Hospital, Bergen, Norway

REFERENCES:
- [Result] Dhayalan D, Tveiten OV, Finnkirk M, Storstein A, Hufthammer KO, Goplen FK, Lund-Johansen M; V-REX Trial investigators. Upfront Radiosurgery vs a Wait-and-Scan Approach for Small- or Medium-Sized Vestibular Schwannoma: The V-REX Randomized Clinical Trial. JAMA. 2023 Aug 1;330(5):421-431. doi: 10.1001/jama.2023.12222. PMID 37526718
- [Derived] Dhayalan D, Tveiten OV, Goplen FK, Finnkirk MK, Storstein AM, Gruner ER, Lund-Johansen M. Comparing the impact of upfront radiosurgery versus expectation in vestibular schwannoma (the V-REX study): protocol for a randomised, observer-blinded, 4-year, parallel-group, single-centre, superiority study. BMJ Open. 2021 Mar 17;11(3):e039396. doi: 10.1136/bmjopen-2020-039396. PMID 33737417